CLINICAL TRIAL: NCT02848716
Title: A Phase III Randomized Study of Pretherapeutic Paraaortic Lymphadenectomy in Women With Locally Advanced Cervical Cancer Dispositioned to Definitive Chemoradiotherapy
Brief Title: Pretherapeutic Paraaortic Lymphadenectomy in Women With Locally Advanced Cervical Cancer Versus Definitive Chemoradiotherapy
Acronym: LiLACs
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study cancelled due to operational difficulties
Sponsor: Muriel POUBLANC (Other)
Responsible Party: Sponsor-Investigator, Muriel POUBLANC, Dr Alejandra MARTINEZ, Institut Claudius Regaud
Organization: Institut Claudius Regaud (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10 GENF 04
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Overall Survival Comparison Between the 2 Arms
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care arm (Active Comparator): Standard chemoradiation based on FluoroDeoxyGlucose-Positon Emission Tomography (FDG-PET) imaging status of the pelvic nodes
  Interventions: Radiation: Standard chemoradiation; Radiation: chemoradiation
- Experimental arm (Experimental): Pretherapeutic paraaortic lymphadenectomy followed by tailored chemoradiation. Pretherapeutic lymphadenectomy will be performed via the laparoscopic extraperitoneal or transperitoneal approach
  Interventions: Procedure: Surgery followed with chemoradiation

INTERVENTIONS:
Procedure: Surgery followed with chemoradiation — Patients with negative paraaortic lymph nodes will be managed with external beam radiotherapy to the pelvis (as defined by the surgical clips applied at the lower limit of the paraaortic node dissection) at a usual dose of 45 Gy. Limited boosts will be indicated individually on clinically involved parametria or pelvic nodes. The external beam radiation therapy will be followed by intracavitary brachytherapy (High Dose Rate (DR), Low DR or Pulse DR) with intent to cure.
  Patients with metastatic disease to paraaortic lymph nodes will receive extended-field external beam radiotherapy followed by intracavitary brachytherapy with intent to cure. Patients who complete both external beam radiation and intracavitary radiotherapy will receive a total dose of 80-90 Gy low-dose equivalent to Point A.
  Concurrent platinum-based chemotherapy (in the 2 sub groups above) will be given with definitive radiation therapy.
  Arms: Experimental arm
Radiation: Standard chemoradiation — patients with negative paraaortic lymph nodes on PET imaging will be managed with external beam radiotherapy to the pelvis at a usual dose of 45 Gy. Limited boosts will be indicated individually on clinically involved parametria or pelvic nodes. The external beam radiation therapy will be followed by intracavitary brachytherapy with intent to cure (HDR, LDR or PDR). Patients who complete both external beam radiation and intracavitary radiotherapy will receive a total dose of 80-90 Gy low-dose equivalent to Point A.
  Concurrent platinum-based chemotherapy will be given with definitive radiation therapy.
  Arms: Standard of care arm
Radiation: chemoradiation
  Arms: Standard of care arm

SUMMARY:
This is an international, prospective, multicenter and randomized phase III study designed to determine if patients with locally advanced cervical cancer have longer overall survivals with pretherapeutic paraaortic surgical staging when compared to radiologic staging.

DETAILED DESCRIPTION:
All eligible patients will be equally randomized between the 2 following treatment groups:

* Standard of care arm: standard chemoradiation (whole pelvis chemoradiation therapy).
* Experimental arm: pretherapeutic paraaortic lymphadenectomy followed by tailored chemoradiation. Pretherapeutic lymphadenectomy will be performed via the laparoscopic extraperitoneal or transperitoneal approach using either traditional laparoscopy or robotically-assisted laparoscopy.

The surgery (extraperitoneal or transperitoneal laparoscopic lymphadenectomy) is considered investigational.

Chemoradiation treatment (with either pelvis or tailored radiation) is considered as standard treatment approved in France for the treatment of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women with clinical stage from 1B2 to 4A cervical squamous cell carcinoma, adenosquamous, or adenocarcinoma.
2. Women with FDG-PET positive or indeterminate pelvic lymph nodes or indeterminate low common iliac nodes (see addendum below) and negative paraaortic nodes.
3. Women with planned treatment of primary definitive chemoradiation therapy.
4. Patient information and written informed consent form signed.
5. Age ≥ 18 years old.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.
7. Life expectancy ≥ 3 months.

Exclusion Criteria:

1. Women with stage 1A or 1B1 cancer.
2. Women with prior radiotherapy to the pelvis or retroperitoneal surgery.
3. Women with neuroendocrine histologies, or histologies other than squamous, adenosquamous or adenocarcinoma.
4. Women with FDG PET positive high common / paraaortic lymph node metastasis confirmed by biopsy (see addendum below).
5. Women who have undergone simple or radical hysterectomy prior to radiotherapy.
6. Women with planned treatment of radiotherapy only (without chemotherapy).
7. Women with planned treatment of palliative radiotherapy.
8. Women with metastatic disease outside of pelvis.
9. Women who have completed treatment for other malignancies (except non-melanomatous skin cancer) < 5 years from their new diagnosis of cervical cancer.
10. Women who are pregnant, women who are likely to be pregnant or are breastfeeding.
11. Women with any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent or compliance to study procedures.
12. Women not affiliated with Social Security System in France.
13. Women deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 10 years
  A Positon Emission Tomography (PET) scan will be obtained at 3 months after completion of chemoradiation therapy. CT scans will be obtained every 6 months for the next three years thereafter. Follow-up surveillance of patients will consist of serial clinical examinations by an oncologist every 3 months for the first 2 years, every 6 months for the next 3 years; then, patients will be followed annually only for collection of their survival data. Patients will come off study at 5 years after completion of initial chemoradiation therapy or at time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Martinez, Dr, Principal Investigator — Institut Claudius Regaud

IPD SHARING:
Plan to Share IPD: Yes
Specific Case Report Form (CRF)